CLINICAL TRIAL: NCT06980038
Title: A Phase 2 Window of Opportunity Trial of Neoadjuvant Agonistic Anti-CD40 Antibody CDX-1140 and Cemiplimab (REGN2810) in AJCC Stage III-IV Head and Neck Cancer Patients Prior to Surgery
Brief Title: Testing Whether Cemiplimab (REGN2810) Plus CDX-1140 Given Prior to Surgery Are Better Than Cemiplimab (REGN2810) Alone in Patients With Stage III-IV Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03539; NCI-2025-03539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10706 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10706 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cutaneous Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Nasal Cavity Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Recurrent Head and Neck Cutaneous Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Nasal Cavity Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Nasopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — Biopsy; Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Cemiplimab) (Active Comparator): Patients receive cemiplimab IV over 30 minutes on day 1. Patients then undergo standard of care surgical resection on day 29-36 and receive standard of care adjuvant therapy. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET during screening and tumor biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Tumor Resection
- Arm II (CDX-1140 and cemiplimab) (Experimental): Patients receive CDX-1140 IV over 90 minutes on day 1 and cemiplimab IV over 30 minutes on day 4. Patients then undergo standard of care surgical resection on day 29-36 and receive standard of care adjuvant therapy. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET during screening and tumor biopsy and blood sample collection throughout the study.
  Interventions: Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Tumor Resection

INTERVENTIONS:
Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140 — Given IV
  Other Names: Agonist CD40 Antibody CDX-1140; Anti-CD40 Agonistic Monoclonal Antibody CDX-1140; CDX 1140; CDX-1140
  Arms: Arm II (CDX-1140 and cemiplimab)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm II (CDX-1140 and cemiplimab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Tumor Resection — Undergo resection surgery

SUMMARY:
This phase II trial compares the effectiveness of cemiplimab with CDX-1140 to cemiplimab without CDX-1140 prior to surgery in treating patients with stage III-IV head and neck cancer. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. CDX-1140 is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Giving cemiplimab with CDX-1140 versus cemiplimab alone before surgery may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed for patients with stage III-IV head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate major pathologic response rate (defined as ≤ 10% of residual viable tumor) of anti-CD40 agonist monoclonal antibody CDX-1140 (CDX-1140) combined with cemiplimab (REGN2810) compared with cemiplimab (REGN2810) alone.

SECONDARY OBJECTIVES:

I. Evaluate the rate of any pathologic response of CDX-1140 in combination with cemiplimab (REGN2810).

II. To evaluate toxicity and tolerability of CDX-1140 and programmed cell death protein 1 (PD-1) blockade combination in neoadjuvant (pre-surgical) setting.

III. To compare gene expression profiles by ribonucleic acid (RNA) sequencing (RNAseq) between CDX-1140 and control groups as well as correlate gene expression with pathologic response.

IV. To evaluate circulating tumor deoxyribonucleic acid (DNA) (ctCNA) as a biomarker of response to neoadjuvant immunotherapy V. To evaluate the pharmacokinetics (PK) of CDX-1140 and cemiplimab (REGN2810) used in combination (arm 2) and the relationship of outcomes to baseline and time-varying clearance of both agents.

EXPLORATORY OBJECTIVES:

I. To evaluate dynamic changes in tumor microenvironment (TME) and circulating immune cell populations.

Ia. To compare dynamic changes in TME while on treatment with subsequent pathologic response in the final specimen.

II. To evaluate changes in circulating plasma cytokines pre and post neoadjuvant immunotherapy with CDX-1140 and cemiplimab (REGN2810).

III. To correlate major pathologic response with the level of programmed cell death ligand 1 (PD-L1) expression.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1. Patients then undergo standard of care surgical resection on day 29-36 and receive standard of care adjuvant therapy. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, positron emission tomography (PET) during screening and tumor biopsy and blood sample collection throughout the study.

ARM II: Patients receive CDX-1140 IV over 90 minutes on day 1 and cemiplimab IV over 30 minutes on day 4. Patients then undergo standard of care surgical resection on day 29-36 and receive standard of care adjuvant therapy. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET during screening and tumor biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at week 9-10, week 18, at 6 months and every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed American Joint Committee on Cancer (AJCC) stage III-IV T0-4, N0-3b, M0 mucosal head and neck squamous cell carcinoma (HNSCC) (oral cavity, oropharynx, larynx, hypopharynx, nasal cavity and skin) that is appropriate for surgical resection. Both previously untreated (primary) and recurrent (salvage) settings will be eligible. Tumors must be accessible to biopsy in clinic (patients with laryngeal, hypopharyngeal, nasal cavity and base of tongue tumors will have endoscopic biopsies)
* For patients with oropharyngeal cancer, only p16-negative (non-human papillomavirus [HPV] related) patients will be eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥ 10 mm (≥ 1 cm) with CT scan, MRI, or calipers by clinical exam
* Age ≥ 18 years. Because no dosing or adverse event (AE) data are currently available on the use of cemiplimab (REGN2810) alone or in combination with CDX-1140 in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Hemoglobin (Hb) ≥ 7 g/dL (transfusion allowed to bring Hb to this level)
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) /alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN
* Creatinine ≤ 1.5 × institutional ULN OR glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Based on its mechanism of action, cemiplimab (REGN2810) can cause fetal harm when administered to a pregnant woman. Animal studies have demonstrated that inhibition of the PD-1/PD-L1 pathway can lead to increased risk of immune-mediated rejection of the developing fetus resulting in fetal death. Women of childbearing potential and men should use effective contraception during treatment with cemiplimab (REGN2810) and for 4 months after the last dose. The reproductive and developmental toxicity of CDX-1140 has not been evaluated. Women of childbearing potential and their partners who receive CDX-1140 must therefore take adequate contraceptive measures
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Active or documented history of autoimmune disease within 2 years before screening
* Prior or planned allogeneic hematopoietic stem cell transplantation (HSCT)
* History of organ transplant that requires use of immunosuppressive medications
* Current or prior use of immunosuppressive medication within 14 days prior to the start of study drug administration. Immunosuppressants may interfere with study drug efficacy
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including cemiplimab (REGN2810). It is unclear how prior exposure to immunotherapy would impact future use of checkpoint inhibitors
* Concurrent use of prednisone (10 mg or more)
* Patients with new pulmonary infiltrates indicative of pneumonitis, history of (non-infectious) pneumonitis/interstitial lung disease, or current pneumonitis/interstitial lung disease, including grade 1 pneumonitis (i.e., asymptomatic, clinical or diagnostic observation only, intervention not indicated)
* Another active malignancy for which the natural history or treatment has potential to interfere with the safety or efficacy assessment of the investigational regimen on this trial
* Patients who have not recovered from AE due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents, such as concurrent chemotherapy, biologic, immunologic or hormonal therapy for cancer treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CDX-1140 or cemiplimab (REGN2810)
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because of the increased risk of immune-mediated rejection of the developing fetus with cemiplimab (REGN2810). Because of the potential for serious adverse reactions in breastfed children, women should not breastfeed during treatment with cemiplimab (REGN2810) and for at least 4 months after the last dose. These risks may also apply to CDX-1140

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-08-21 (Estimated); Primary Completion 2027-11-24 (Estimated); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | From the time of their first treatment with CDX-1140 and/or cemiplimab (REGN2810), up to 2 years
  Will be assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Descriptive statistics will be used.
Major pathologic response | Up to 2 years
  Defined as ≤ 10% of viable tumor area relative to total tumor area.

SECONDARY OUTCOMES:
Acute incidence of adverse events | From the time of their first treatment with CDX-1140 and/or cemiplimab (REGN2810), up to 2 years
  Will be assessed using NCI CTCAE version 5.0. Descriptive statistics will be used.
Late incidence of adverse events | From the time of their first treatment with CDX-1140 and/or cemiplimab (REGN2810), up to 2 years
  Will be assessed using NCI CTCAE version 5.0. Descriptive statistics will be used.
Quantitative pathologic response | Up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes.
Tumor infiltrating immune populations | Up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes.
Serum cytokines levels | Up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes.
Circulating tumor deoxyribonucleic acid (ctDNA) levels | Up to 2 years
  Two-sample t-test, Mann-Whitney U test, or log rank test will be used where appropriate to analyze the correlation between efficacy outcomes. Will also compare ctDNA levels between the two arms and between responders and non-responders using a Student's t-test.
Gene expression levels | Day 3 and day 29-36
  Will be assessed using DEseq2, and will also be compared between treatment arms and between those with and without achieving pathologic response.
Gene set enrichment | Up to 2 years
  Gene set statistics will be run with fgsea using MSigDb61 pathways annotated in the HALLMARK databases.
Pharmacokinetic (PK) parameters | Up to study completion
  Including clearance and area-under-the-curve, will be calculated for cemiplimab (REGN2810) and CDX-1140 in combination. Impact of baseline and time-varying clearance of cemiplimab (REGN2810) and CDX-1140 in combination will be correlated to efficacy data and AEs to evaluate any PK-related efficacy or toxicity relationship. Also, comparison of observed cemiplimab (REGN2810) PK with historical data will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Matin Imanguli, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (1):
- JHU Sidney Kimmel Comprehensive Cancer Center LAO, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm